CLINICAL TRIAL: NCT02638610
Title: Assessment of Changes of Periocular Skin Sensation Following Eyelid and Ocular Surface Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC 0110-15
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Blepharoptosis; Blepharochalasis, Superior; Ectropion; Entropion
MeSH Terms: conditions — Blepharoptosis; Blepharochalasis, Superior; Ectropion; Entropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensation measurement (Experimental): patients with eyelid pathology going through eyelid surgery.
  Interventions: Device: Cochet-Bonnet aesthesiometer

INTERVENTIONS:
Device: Cochet-Bonnet aesthesiometer — The eyelid's sensation will be assessed at 6 points of the eyelid using the Cochet-Bonnet aesthesiometer (Luneau Ophtalmologie, Paris, France). Measurements will take place before surgery, and two weeks, three months and six months after surgery.
  This instrument contains a 6 centimeters long, retractable, flexible monofilament. For any given length, when applied perpendicularly to a test surface, the filament will exert a precise pressure before visibly bending. The filament's length inversely corresponds to the pressure exerted by the aesthesiometer such that the shorter the filament length, the more pressure it exerts on the test surface.

SUMMARY:
The aim of the study: Assessment of Changes of Periocular Skin Sensation Following Eyelid and Ocular Surface Surgeries.

Study design: an interventional study that will be conducted at the ophthalmology department, Meir hospital, Kfar Saba, Israel.

the study will include 60 healthy patients, at the ages of 40-80, which are candidates for eyelid surgery: blepharoptosis repair, blepharoplasty, ectropion repair and entropion repair.

The patients will be recruited from Meir's ophthalmology outpatient clinic. Each patient will undergo a full ophthalmologic examination including relevant assessment of the specific eyelid pathology.

The eyelid's sensation will be assessed at 6 points of the eyelid using the Cochet-Bonnet filament-type aesthesiometer (Luneau Ophtalmologie, Paris, France). Measurements will take place before surgery, and two weeks, three months and six months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give consent
* Eyelid pathology: blepharoptosis, blepharochalasis, ectropion or entropion, with no additional eyelid pathology

Exclusion Criteria:

* Children and pregnant women
* Previous eyelid surgery
* A systemic disease influencing eyelid position
* Any neurologic disease
* Previous facial herpetic infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Changes of periocular skin sensation following eyelid and ocular surface surgeries (expressed in the length of the aesthesiometer's filament in centimeters). | 6 months

IPD SHARING:
Plan to Share IPD: Undecided